CLINICAL TRIAL: NCT04445727
Title: Efficacy of Vitamin C Supplement Addiction vs. High-speed Spinal Manipulation to Routine Physiotherapy Treatment in Lateral Epicondylitis
Brief Title: Efficacy of Vitamin C Supplement vs Spinal Manipulation to Treatment in Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Pablo Federico Scillone Tessore, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PScillone
Record Dates: First submitted 2020-06-14; First posted 2020-06-24 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: Acid, Ascorbic; Transcutaneous Electric Nerve Stimulation; Spinal Manipulation; Musculoskeletal Manipulations
MeSH Terms: conditions — Tennis Elbow; Heartburn | interventions — Ascorbic Acid; Transcutaneous Electric Nerve Stimulation; Musculoskeletal Manipulations; Manipulation, Spinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- vitamin c (Experimental): daily dose of 1000 mg vitamin c in order to regenerate collagen
  Interventions: Combination Product: Transcutaneous electrical nerve stimulation (TENS)
- spinal manipulation (Experimental): Spinal manipulation in cervical and dorsal with high speed and short amplitude techniques
  Interventions: Combination Product: Transcutaneous electrical nerve stimulation (TENS)
- Transcutaneous electrical nerve stimulation (TENS) (Experimental): electrotherapy for an analgesic purpose
  Interventions: Combination Product: Vitamin C; Combination Product: spinal manipulation
- manual therapy (Experimental): manual muscle treatment for epicondyl musculature
  Interventions: Combination Product: Vitamin C; Combination Product: spinal manipulation; Combination Product: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Combination Product: Vitamin C — Will apply 1000mg of vitamin C, TENS and manual therapy. One session will be held per week for 6 weeks.
  Other Names: tens; manual therapy
  Arms: Transcutaneous electrical nerve stimulation (TENS); manual therapy
Combination Product: spinal manipulation — Applied spinal manipulations, tens and manual therapy.One session will be held per week for 6 weeks.
  Other Names: tens; manual therapy
  Arms: Transcutaneous electrical nerve stimulation (TENS); manual therapy
Combination Product: Transcutaneous electrical nerve stimulation (TENS) — Received a manual therapy intervention and Tens. one session will be held per week for 6 weeks.
  Other Names: manual therapy
  Arms: manual therapy; spinal manipulation; vitamin c

SUMMARY:
A randomized clinical trial will be conducted. 130 subjects diagnosed with lateral epicondylitis will be studied. 3 intervention groups will be formed. Experimental group 1 will receive a 1000mg daily vitamin C supplement along with the usual practice of manual therapy and TENS. Group 2 will undergo high-speed vertebral manipulations along with manual therapy and TENS. In group 3 or control, manual therapy and transcutaneous electrotherapy (TENS) will be applied. All groups will receive the same manual therapy program and TENS, one session per week for 6 consecutive weeks. Data analysis: The data will be entered in the SPSS statistical package (version 21.0) for analysis). Statistical analysis will be performed with a 95% confidence interval, meaning that those whose P is <0.05 will be considered significant values.

DETAILED DESCRIPTION:
The 130 subjects will be randomized into 3 groups: Experimental group 1 will receive a supplement of vitamin C (ascorbic complex) of the Bonusan brand, a daily dose of 1000mg should be consumed along with the usual practice of manual therapy and TENS. This group will maintain the daily intake of vitamin C for the 6 weeks that the treatment lasts, they will be informed of the possible side effects of adaptation to the supplement, such as, for example, diarrhea since excess vitamin C, in the case if there is, it lodges in the large intestine, which attracts fluid and produces osmotic diarrhea. This group will have direct communication with the doctor who collaborates in this investigation for any situation, query or unwanted symptom. Vitamin C has been used in other degenerative-type pathologies of collagen tissue such as Achilles tendinopathies and supraspinatus musculature. The investigators have also found references to the effect of vitamin C as pain treatment. Group 2 will undergo high-speed vertebral manipulations along with manual therapy and TENS. Vertebral manipulations would seek a reflexogenic effect through the sympathetic nerve pathway of the lower cervical ganglion. The transcutaneous TENS-type stimulation is evidenced to have an analgesic effect using self-adhesive patches placed longitudinally at the myo-junction. tendon with a size of 50X50 mm, a frequency of 100 Hz and a pulse duration of 200μs for 25 minutes. Both the vertebral manipulation intervention and the TENS placement will be performed by a professional health physiotherapist with 27 years of clinical experience in the application of the aforementioned techniques.

In group 3 or control, manual therapy and transcutaneous electrotherapy (TENS) will be applied. All groups will receive the same manual therapy program and TENS, one session per week for 6 consecutive weeks.

All the aforementioned interventions will be included in a 45 minute session for the 3 groups alike. They will be in charge of a highly qualified physiotherapist for all the therapies when carrying out which expresses his consent for the study in. Said professional uses all these therapies in consultation daily.

8 The aforementioned therapies can generate some adverse effects that the participants should be aware of and that is reflected in the informed consent that they must complete before the start of the evaluation and the interventions. In the first place, in the TENS, no bibliography has been found that warns of any unwanted effect, which it can refer to is an increase in skin tone under the patch due to the local effect and heat conduction of the same. which should disappear within 30 minutes after application.

In high-speed vertebral manipulation in the cervical region, in 6% of cases, post-manipulation dizziness may occur due to the local vascular change that occurs . The vitamin C supplement can produce some type of heartburn diarrhea, especially in the first days of taking, since this vitamin is absorbed in the intestine .

Alterations at the elbow can cause pain and functional limitation. To quantify these effects, there are different measurement scales. The evaluation to quantify the pain will be carried out with the numerical pain scale (0-10). The Disabilities of the Arm Shoulder and Hand (DASH) questionnaire will be used to determine the functionality of the upper limb, the Shoulder Pain and Disability Index SPADI will be used to assess shoulder function, Global perception of change will also be evaluated, Global Rating of Change Scale (GROC) a 15-point scale where -7 indicates much worse than before, 0 the same as before and +7 much better than before . Finally, the pressure pain threshold (PDU) will be evaluated using a digital algometer .

Measurement variables will be analyzed before treatment, after it, and at 3 and 6 months after the last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Elbow pain patients medically diagnosed with epicondylitis by ultrasound of more than 4 weeks of evolution.
* Age between 35 and 55 years (both inclusive).
* Have signed the informed consent.

Exclusion Criteria:

* Have received corticosteroid infiltrations in the previous 3 months. Having received physical therapy treatment for the same reason in last 3 months.
* Bilateral symptoms.
* Fibromyalgia syndrome.
* Previous trauma to the upper limb.
* Fractures or prior dislocation of the shoulder or elbow.
* Previous surgeries on the shoulder or elbow.
* Psychiatric treatment.
* Cognitive deficit.
* Owning defibrillator or pacemaker.
* Acute infectious diseases.
* Uncontrolled systemic pathologies (heart disease, pacemaker, coagulation disorders).
* Pregnant women.
* History of rheumatic disease affecting the elbow such as rheumatoid arthritis, gout, reflex sympathetic dystrophy, plaque psoriasis. • Oncological processes.
* Aversion or fear of the application of currents.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-03-11 (Estimated)

PRIMARY OUTCOMES:
Pain will be measured using an analog visual Scale | 6 weeks
  For this, patients will be indicated how they should complete the scale, providing a numerical value from 0 to 10, being 10 0 no pain, and 10 the most severe or intense pain. The numerical pain scale is a simple, solid, sensitive and reproducible instrument, useful for reassessing patient pain

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Scale | 6 weeks
  The questionnaire will consist of 30 questions about their symptoms and the ability to carry out certain activities and has been validated in Spanish. The patient should answer the questions by circling the number that best describes their condition during the past week. Each item will be answered on a scale from 1 to 5, where 1 indicates that it has no difficulty executing, has no symptoms or impact, and 5 indicates that it cannot be performed, that it has very severe symptoms and a strong impact.

OTHER OUTCOMES:
Global Rating of Change Scale | 6 weeks
  The 15-point improvement self-perception scale (GROC) will be used, consisting of a 15-point Likert scale ranging from a rating of 0 to +7 (I am much better) or -7 (I am much worse).
  eleven The descriptors of improvement range from +1 to +7, and those of worsening from -1 to -7. A value of +5 has been shown to be indicative of moderate clinical improvement, while a value of +6 or +7 suggests high clinical improvement.
Algometry | 6 weeks
  Pressure pain threshold will be analyzed, defined as the minimum amount of pressure applied to produce pain

CONTACTS AND LOCATIONS:
Overall Officials: Ana I de la Llave Rincón, Study Director — Universidad Rey Juan Carlos; José J Arias Buría, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Pablo Federico Scillone Tessore, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Notarnicola A, Pesce V, Vicenti G, Tafuri S, Forcignano M, Moretti B. SWAAT study: extracorporeal shock wave therapy and arginine supplementation and other nutraceuticals for insertional Achilles tendinopathy. Adv Ther. 2012 Sep;29(9):799-814. doi: 10.1007/s12325-012-0046-4. Epub 2012 Aug 24. PMID 22923162
- [Result] Leijn E, Monnens LA, Cornelissen EA. Intravenous iron supplementation in children on hemodialysis. J Nephrol. 2004 May-Jun;17(3):423-6. PMID 15365964
- [Result] Passerieux E, Hayot M, Jaussent A, Carnac G, Gouzi F, Pillard F, Picot MC, Bocker K, Hugon G, Pincemail J, Defraigne JO, Verrips T, Mercier J, Laoudj-Chenivesse D. Effects of vitamin C, vitamin E, zinc gluconate, and selenomethionine supplementation on muscle function and oxidative stress biomarkers in patients with facioscapulohumeral dystrophy: a double-blind randomized controlled clinical trial. Free Radic Biol Med. 2015 Apr;81:158-69. doi: 10.1016/j.freeradbiomed.2014.09.014. Epub 2014 Sep 20. PMID 25246239
- [Result] Malek Mahdavi A, Mahdavi R, Kolahi S, Zemestani M, Vatankhah AM. L-Carnitine supplementation improved clinical status without changing oxidative stress and lipid profile in women with knee osteoarthritis. Nutr Res. 2015 Aug;35(8):707-15. doi: 10.1016/j.nutres.2015.06.003. Epub 2015 Jun 16. PMID 26149189
- [Result] Lee GW, Yang HS, Yeom JS, Ahn MW. The Efficacy of Vitamin C on Postoperative Outcomes after Posterior Lumbar Interbody Fusion: A Randomized, Placebo-Controlled Trial. Clin Orthop Surg. 2017 Sep;9(3):317-324. doi: 10.4055/cios.2017.9.3.317. Epub 2017 Aug 4. PMID 28861199
- [Result] Coombes BK, Bisset L, Vicenzino B. Bilateral cervical dysfunction in patients with unilateral lateral epicondylalgia without concomitant cervical or upper limb symptoms: a cross-sectional case-control study. J Manipulative Physiol Ther. 2014 Feb;37(2):79-86. doi: 10.1016/j.jmpt.2013.12.005. Epub 2013 Dec 28. PMID 24378321
- [Result] Fernandez-Carnero J, Fernandez-de-las-Penas C, Cleland JA. Immediate hypoalgesic and motor effects after a single cervical spine manipulation in subjects with lateral epicondylalgia. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):675-81. doi: 10.1016/j.jmpt.2008.10.005. PMID 19028251
- Available data/document: Clinical Study Report: vitamin c — http://www.bonusan.es/vademecum/vitamina_c1000_complejo_de_ascorbatos.html